CLINICAL TRIAL: NCT00125242
Title: Word-Retrieval for Aphasia: Facilitation of Generalization
Brief Title: Word-Retrieval Treatment for Aphasia: Semantic Feature Analysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C3826-R
Record Dates: First submitted 2005-07-27; First posted 2005-07-29 (Estimated); Results first posted 2014-12-24 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Aphasia; Language Disorders; Speech Disorders
Keywords: Aphasia; Language therapy; Rehabilitation of speech and language disorders; Speech-language pathology
MeSH Terms: conditions — Aphasia; Language Disorders; Speech Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Semantic Feature Analysis (SFA) (Experimental): Word retrieval treatment for aphasia.
  Interventions: Behavioral: Semantic Feature Analysis (SFA)Training
- Participants for Stimuli Development (No Intervention): Non-brain-injured participants provided data for development of treatment stimuli.

INTERVENTIONS:
Behavioral: Semantic Feature Analysis (SFA)Training — SFA entails having the speech-language pathologist (SLP) guide the participant through generation of pertinent semantic features for pictured treatment items (e.g., category membership, physical description, location of item in context, personal associations, action associated with item). For some participants, treatment items were grouped according to typicality of category membership (e.g,, a robin-typical bird and penguin-atypical bird). Training of atypical items may stimulate a broader semantic activation of the category and thus, may promote greater generalization. Treatment was applied sequentially to sets of items in the context of single-subject, multiple baseline designs. In this way, replication of treatment effects could be evaluated within and across participants. Treatment was administered by certified SLPs three times per week until prescribed accuracy levels were met during nontreatment probes or a maximum number of treatment sessions was completed.
  Arms: Semantic Feature Analysis (SFA)

SUMMARY:
The purpose of this investigation is to further develop and test a treatment for word-finding problems in aphasia. The treatment is designed to strengthen meaning associations within categories of words (e.g., animals, tools, fruits). The treatment is also designed to be used as a search strategy in instances of word-finding difficulty. The study was devised to evaluate the extent to which treatment increases the ability to recall trained, as well as untrained, words.

DETAILED DESCRIPTION:
The purpose of the proposed research is to examine the effects of a semantically-oriented treatment on word retrieval in persons with aphasia. The planned investigations are designed to further the development of semantic feature training so that it may serve as not only a mechanism for improving disrupted lexical semantic processing, but also as a compensatory strategy during word retrieval failures. The proposed research will also address the issue of exemplar typicality (Kiran & Thompson, 2003) by examining the effects of training typical versus atypical exemplars of various categories with individuals with different types of aphasia. A series of 24 single subject experimental designs will be conducted in the context of a group design to address the following experimental questions:

* Will training atypical examples of living and artifact noun categories using semantic feature training result in a significantly different outcome* than training typical examples of living and artifact noun categories?
* Will training of one category of nouns using semantic feature training result in improved retrieval of untrained categories of nouns?
* Will effects of semantic feature training vary across aphasia types?
* Will semantic feature training result in increased production of content during discourse?
* Will generalization to untrained typical examples vary across generalization lists that are repeatedly exposed and those that are limited in exposure? (i.e., Does repeated exposure appear to contribute to generalization?)

  * Outcome measure will reflect acquisition, response generalization within category, and response generalization across category effects of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Wernicke's, Broca's, or Conduction aphasia with significant word-retrieval deficits
* At least 6 months post-onset of single, left-hemisphere stroke
* Minimum of high-school education
* Visual and auditory acuity sufficient for experimental tasks
* Nonverbal intelligence within normal limits

Exclusion Criteria:

* Diagnosed mental illness other than depression
* Neurological condition other than that which resulted in aphasia
* History of alcohol or substance abuse
* Non-native English speaker
* Premorbid history of speech/language disorder

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2005-07; Primary Completion 2009-02 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie L. Wambaugh, PhD, Principal Investigator — VA Salt Lake City Health Care System, Salt Lake City
Locations (1):
- VA Salt Lake City Health Care System, Salt Lake City, Salt Lake City, Utah, United States

REFERENCES:
- [Result] Wambaugh JL, Mauszycki S, Cameron R, Wright S, Nessler C. Semantic feature analysis: incorporating typicality treatment and mediating strategy training to promote generalization. Am J Speech Lang Pathol. 2013 May;22(2):S334-69. doi: 10.1044/1058-0360(2013/12-0070). PMID 23695909
- [Result] Wambaugh JL, Mauszycki S, Wright S. Semantic feature analysis: Application to confrontation naming of actions in aphasia. Aphasiology. 2013 Oct 28; 28(1):DOI:10.1080/02687038.2013.845739.

RESULTS

PARTICIPANT FLOW:
Groups:
- Non Treatment Stimuli Development Participants: Non-brain-injured participants who were enrolled for the purpose of stimuli development
- SFA Treatment Participants: Stroke survivors who received experimental therapy
Period: Overall Study
Arm/Group | Non Treatment Stimuli Development Participants | SFA Treatment Participants
Started | 94 | 16
Completed | 87 | 14
Not Completed | 7 | 2
Not completed — did not qualify | 7 | 2

BASELINE CHARACTERISTICS:
Population: SFA Treatment Participants = Stroke survivors with chronic aphasia. Non Treatment Stimuli Development Participants = non-brain-damaged persons who were enrolled for purposes of stimuli development.
Groups:
- SFA Treatment Participants: Semantic Feature Analysis (SFA) is a word-retrieval treatment for aphasia. SFA entails having the speech-language pathologist (SLP) guide the participant through generation of pertinent semantic features for pictured treatment items (e.g., category membership, physical description, location of item in context, personal associations, associated actions). For some participants, treatment items were grouped by typicality of category membership (e.g, robin-typical bird and penguin-atypical bird). Training of atypical items may stimulate a broader semantic activation of the category and thus, may promote greater generalization. Treatment was applied sequentially to sets of items in single-subject, multiple baseline designs. Thus, replication of treatment effects could be evaluated within and across participants. Treatment was administered by SLPs three times per week until prescribed accuracy levels were met during probes or a maximum number of treatment sessions was completed.
- Non Treatment Stimuli Development Participants: Participants for stimuli development provided normative data for stimuli development. e.g., Treatment items were grouped according to typicality of category membership (apple - typical fruit; coconut - atypical fruit). These participants provided the reponses that served as the basis for classifying/organizing stimuli. Because data from this group were used only for the purposes of stimuli development, no findings are reported for this group. See Cameron, R.M., Wambaugh, J.L., & Mauszycki, S. (2008). Effects of age, gender and education on semantic fluency for living and artifact categories. Aphasiology, 22(7/8), 790-801, doi: 10.1080/02687030701818018 for related findings.
- Total: Total of all reporting groups
Arm/Group | SFA Treatment Participants | Non Treatment Stimuli Development Participants | Total
Number analyzed (Participants) | 16 | 94 | 110
Age, Customized [Number; unit: participants]
  21-80 Years | 16 | 94 | 110
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 47 | 51
  Male | 12 | 47 | 59

OUTCOME MEASURES:

1. Primary Outcome: Word Retrieval Accuracy
Description: Accuracy of naming of pictured treated and untreated items was assessed in probes conducted separate from treatment. Probes were conducted repeatedly throughout the study, from baseline (prior to treatment) to follow-up (6 weeks following treatment). All naming responses were scored using a 0-10 scale reflecting promptness and presence of errors; scores of 8-10 received an "accuate" score and scores of 0-7 received an "inaccurate" score. A percentage accuracy score was calculated for each experimental set of items for every probe session. Baseline probe scores were compared to end of treatment and follow-up probe scores to obtain individual effect sizes for each experimental list of items for each participant (i.e., several effect sizes were calculated for each participant). All effect sizes were utlized to obtain an average effect size for each participant; these averages were then utlized to obtain a group average.
Time Frame: End of treatment and at 6 weeks post treatment
Population: SFA Treatment Participants were stroke-survivors with chronic aphasia who had significant word retrieval difficulties. Non Treatment Stimuli Development Participants were only enrolled in the study to provide data for the development of treatment stimuli. As such, they were not assessed for the outcome measure.
Measure: Mean (Standard Deviation); unit: d-index (effect size)
Units Other Than Participants: participant effect sizes
Groups:
- SFA Treatment Participants: Stroke survivors received Semantic Feature Analysis for the treatment of word-retrieval deficits. Each SFA treatment participant received word-retrieval therapy applied sequentially to experimental lists of items. Effect sizes were calculated for each participant for each list. An average effect size was calculated for each participant and an overall average was determined for all participants as a group.
Arm/Group | SFA Treatment Participants
Number analyzed (Participants) | 13
Number analyzed (participant effect sizes) | 68
d-index (effect size) | 7.15 (3.1)
Statistical Analysis 1: Comparison: SFA Treatment Participants; Effect sizes were calculated - this is a comparison of perfomance in baseline (repeated measurements prior to treatment) relative to peformance following treatment; Test type: Superiority or Other; effect size = 7.15, Standard Deviation 3.1 — the reported effect size is a d-index value

ADVERSE EVENTS:
Time Frame: 3 years
Groups:
- SFA Treatment Participants: Stroke-survivors who received Semantic Feature Analysis therapy for aphasic word-retrieval deficits
  Semantic Feature Training: The treatment is designed to stimulate the semantic feature network so that it may serve as not only a mechanism for improving disrupted lexical semantic processing, but also as a compensatory strategy during word retrieval failures.
- NonTreatment Stimuli Development Participants: Non-brain-injured participants who were utilized to develop treatment stimuli.
Arm/Group | SFA Treatment Participants | NonTreatment Stimuli Development Participants
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/94
Other Adverse Events (participants affected / at risk) | 0/16 | 0/94

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes